CLINICAL TRIAL: NCT01386021
Title: Single Center Evaluation of CryoVein Saphenous Vein Allografts for Coronary Artery Bypass Grafting
Brief Title: Saphenous Vein Allografts for Coronary Bypass
Status: Completed | Type: Observational
Sponsor: CryoLife, Inc. (Industry)
Responsible Party: Sponsor
Organization: CryoLife (Unknown)
Other Study IDs: AVG1101.001-M
Record Dates: First submitted 2011-06-29; First posted 2011-06-30 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Coronary Artery Disease; Occlusion of Artery
Keywords: allograft; coronary; patency; morbidity
MeSH Terms: conditions — Coronary Artery Disease; Arterial Occlusive Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prior recipients of allografts for CABG

SUMMARY:
The primary objective of this observational study is to evaluate the function (patency) of cryopreserved saphenous vein allografts used as coronary artery bypass grafts (CABG) for patients with occlusive coronary artery disease.

DETAILED DESCRIPTION:
This Study is designed as a combination retrospective/prospective single center study in which all patients will be eligible for enrollment based on having a previous implant of CryoVein Saphenous Vein for CABG during the 2008-2010 time frame. A comprehensive chart review of former and previously implanted allograft patients will be performed for the retrospective portion of this Study. An effort will be made to include all patients from this site. Eligible patients will be consented into the Study for a single, prospective, observational imaging evaluation of their bypass conduits.

ELIGIBILITY:
Inclusion Criteria:

* Any patient implanted with a CryoVein saphenous vein allograft for CABG during 2008 - 2010 time frame.
* Patients > 18 years of age at implant.

Exclusion Criteria:

• Patients < 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having a previous implant of CryoVein Saphenous Vein allografts for CABG between 2008 - 2010, at a single instituion
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Graft Patency | 1 to 3 years as defined by the date of their incident operation (CABG surgery).

SECONDARY OUTCOMES:
Morbidity | 1 to 3 years defined by the date of their incident operation (CABG surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Valavanur A Subramanian, M.D., Principal Investigator
Locations (1):
- Lenox Hill Hospital, New York, New York, United States